CLINICAL TRIAL: NCT06831435
Title: Effectiveness of Digital Cognitive Behavioral Therapy for the Treatment of Depression: a Real-world Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University (Other)
Responsible Party: Principal Investigator, Weihua Yue, Professor, Peking University Sixth Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-83
Record Dates: First submitted 2025-02-12; First posted 2025-02-18 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Depression; Bipolar Affective Disorder; Schizophenia Disorder; Psychiatric &Amp;or Mood Disorder
Keywords: i-CBT; a real-world study
MeSH Terms: conditions — Depression; Bipolar Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- i-CBT group (Experimental): i-CBT combined with conventional drug treatment
  Interventions: Device: a digital product based on CBT

INTERVENTIONS:
Device: a digital product based on CBT — The digital cognitive behavioral therapy in this study is conducted based on a self-developed mobile applet. The therapy is developed by psychotherapists, which is conducted for a total of 8 weeks, with weekly sessions including Al-guided course work and homework.

SUMMARY:
The project proposes to develop a digital product based on cognitive behavioral therapy for the assisted treatment of depression. The digital cognitive behavioral therapy in this study is conducted based on a self-developed mobile applet. The therapy is developed by psychotherapists, which is conducted for a total of 8 weeks, with weekly sessions including AI-guided course work and homework. This study aims to evaluate the therapeutic effects of CBT-based digital products for depression in patients through a real-world study, and to explore its genetic and neuroimaging mechanisms.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 14-60 years (including 14 and 60), no gender restriction;
2. HAMD >= 14;
3. Written informed consent obtained from the patient; written informed consent obtained from the guardian for minors.

Exclusion Criteria:

* Persons with severe suicidal tendencies (item 10 of the MADRS scale ≥ 5).

Ages: 14 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 325 (Estimated)
Dates: Start 2024-11-13 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in Hamilton Depression Rating Scale (HAMD) | Week 4 and 8 of treatment duration
  The outcome is assessed by 17-item Hamilton Depression Rating Scale (HAMD-17) Scale. Total HAMD scores range from 0 to 52, with higher scores indicating more severe depressive symptoms. The change of HAMD from baseline to 8-week (after intervention) was used as the primary outcome.

SECONDARY OUTCOMES:
Change from baseline in Montgomery-Asberg Depression Rating Scale (MADRS) | Week 4 and 8 of treatment duration
  The outcome is assessed by Montgomery-Asberg Depression Rating Scale (MADRS). Total MADRS score ranges from 0 to 60, with higher scores indicating greater severity of depression. The change of MADRS from baseline to 8-week (after intervention) was used.
Change from baseline in Positive and Negative Syndrome Scale (PANSS) | Week 4 and 8 of treatment duration
  The outcome is assessed by the Positive and Negative Syndrome Scale (PANSS). The PANSS consists of 30 items, divided into three subscales: Positive Symptoms (7 items), Negative Symptoms (7 items), and General Psychopathology (16 items). Each item is rated on a 7-point scale from 1 (absent) to 7 (extreme), with higher scores indicating more severe symptoms. The total PANSS score ranges from 30 to 210, with higher scores reflecting greater symptom severity.
Response to treatment | Week 4 and 8 of treatment duration
  Reduction rate of Hamilton Depression Scale (HAMD-17) or Montgomery-Asberg Depression Rating Scale (MADRS) score ≥50% was recognized as response to treatment.
Clinical Global Impression-Severity of Illness (CGI-S) | Week 4 and 8 of treatment duration
  The outcome was assessed by the Clinical Global Impression-Severity of Illness (CGI-S) scale. It is rated on a 7-point scale. Higher scores indicate more severe symptoms.
Change from baseline in Hamilton Anxiety Rating Scale (HAMA) | Week 4 and 8 of treatment duration
  The outcome is assessed by 14-item Hamilton Anxiety Scale (HAMA). Total score ranges from 0 to 56, with higher scores indicating greater severity of anxiety. The change of HAMA from baseline to 8-week (after intervention) was used.
Change from baseline in Ruminative Responses Scale (RRS) | Week 4 and 8 of treatment duration
  This outcome is assessed by Ruminative Responses Scale (RRS). Total score ranges from 22 to 88, with higher scores indicating greater severity of rumination. The change of RRS from baseline to 8-week (after intervention) was used.
Change from baseline in Pittsburgh Sleep Quality Index (PSQI) | Week 4 and 8 of treatment duration
  This outcome is assessed by Pittsburgh Sleep Quality Index (PSQI). Total score ranges from 0 to 21, with higher scores indicating greater severity of sleep problems. The change of PSQI from baseline to 8-week (after intervention) was used.
Change from baseline in Connor-Davidson Resilience Scale (CD-RISC) | Week 4 and 8 of treatment duration
  This outcome is assessed by Connor-Davidson Resilience Scale (CD-RISC). Total score ranges from 0 to 100, with higher scores indicating greater resilience. The change of CD-RISC from baseline to 8-week (after intervention) was used.
Change from baseline in Thinc-Integrated Tool(THINC-it) | Week 8 of treatment duration
  Cognitive function was assessed by Thinc-Integrated Tool(THINC-it) using digital device. The change of THINC-it from baseline to 8-week (after intervention) was used.
Mood Disorder Questionnaire (MDQ) | Week 4 and 8 of treatment duration
  This outcome is assessed by Mood Disorder Questionnaire (MDQ), which is used to assess the positive symptom of bipolar. A positive screening for bipolar disorder is determined when there are ≥7 of the 13 screening symptoms present, at least one "yes" response in the second section indicating the co-occurrence of several symptoms, and a severity level of "moderate" or "serious problem" in the third section.
Rating Scale for Side Effects（SERS） | Week 4 and 8 of treatment duration
  This outcome is assessed by Rating Scale for Side Effects (SERS), which assess 13 side-effects. Total score ranges from 13 to 52, with higher scores indicating more side-effects.
Client Satisfaction Questionnaire-3 （CSQ-3) | Week 8 of treatment duration
  User's satisfaction was assessed by Client Satisfaction Questionnaire-3 （CSQ-3). Total score ranges from 3 to 12. with higher scores indicating greater satisfaction.
Change from baseline in Young Mania Rating Scale (YMRS) | Week 4 and 8 of treatment duration
  The outcome is assessed by the Young Mania Rating Scale (YMRS). The YMRS consists of 11 items that assess the severity of manic symptoms, including mood, speech, motor activity, sexual interest, sleep, and other behaviors. Each item is rated on a scale from 0 to 4, with higher scores indicating greater severity of manic symptoms. The total YMRS score can range from 0 to 44, with higher scores reflecting more severe mania.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University Sixth Hostipal, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No